CLINICAL TRIAL: NCT06528301
Title: A Phase 1, Multicenter, Open-label Study of UB-VV111 in Combination With Rapamycin in Relapsed/Refractory (R/R) CD19+ B-cell Malignancies
Brief Title: A Phase 1 Study of UB-VV111 With and Without Rapamycin in Relapsed/Refractory CD19+ B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Umoja Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UB-VV111-01
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Non-Hodgkin (NHL); Lymphoma, Large B-Cell, Diffuse (DLBCL); Chronic Lymphocytic Leukemia (CLL)
Keywords: CAR T; CD19; chimeric antigen receptor
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UB-VV111 (Experimental): A single dose of UB-VV111 will be administered.
  Interventions: Genetic: UB-VV111
- UB-VV111 + rapamycin (Experimental): A single dose of UB-VV111 will be administered followed by treatment with rapamycin.
  Interventions: Genetic: UB-VV111; Drug: rapamycin

INTERVENTIONS:
Genetic: UB-VV111 — UB-VV111 is a gene therapy that generates CD19 CAR T cells in the body.
Drug: rapamycin — Rapamycin is an FDA-approved drug.
  Other Names: Rapamune, sirolimus
  Arms: UB-VV111 + rapamycin

SUMMARY:
This study is a Phase 1 dose-escalation and dose-confirmation study to evaluate the safety and antitumor activity of UB-VV111. The study will enroll patients with relapsed/refractory large B-cell lymphoma (LBCL) and chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Provides voluntary written informed consent
3. Relapsed or refractory large B-cell lymphoma (LBCL) or chronic lymphocytic leukemia (CLL)
4. Measurable disease according to Lugano 2014 criteria (LBCL) or iwCLL 2018 (CLL).
5. No serious concomitant diseases or active/uncontrolled infections
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Adequate organ function
8. Patients who have previously received CD19-directed therapy must have biopsy confirming CD19 expression following completion of prior CD19-directed therapy.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding
2. Current isolated central nervous system (CNS) involvement
3. Prior allogeneic bone marrow transplant, gene therapy, or adoptive cell transfer (except CAR T-cell therapy in CAR T-exposed subjects)
4. History of or active human immunodeficiency virus (HIV)
5. Active hepatitis B or C
6. Systemic autoimmune or immunodeficiency diseases, except for well-controlled Type I diabetes or thyroid disease
7. Ongoing CNS disease that would preclude neurologic assessment
8. Uncontrolled angina or other acute heart disease
9. Currently receiving treatment in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with common adverse events (AEs) | Up to 2 years after UB-VV111 administration
  Percentage of participants with commonly reported AEs overall and by severity

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years after UB-VV111 administration
  Percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Garcia, MD, Study Director — Umoja Biopharma
Locations (8):
- United States (6):
  - City of Hope, Duarte, California
  - The David and Etta Jonas Center for Cellular Therapy, Chicago, Illinois
  - Washington University School of Medicine/Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Cincinnatti Medical Center, Cincinnati, Ohio
  - Fred Hutch Cancer Center, Seattle, Washington
- Australia (2):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria

IPD SHARING:
Plan to Share IPD: No